CLINICAL TRIAL: NCT05744700
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Determine the Safety and Tolerability of Microbial Inulinase
Brief Title: Safety and Tolerability Trial of Microbial Inulinase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIO-CAT, Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B03-22-01-T0037; BCCT-AB-0009 (Other: BIO-CAT, Inc.)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Digestive Health; Gastrointestinal Health
MeSH Terms: interventions — inulinase; beta-Fructofuranosidase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inulinase (Active Comparator): Total 2,000 INU inulinase per day for 28 days
  Interventions: Dietary Supplement: Inulinase
- Placebo (Placebo Comparator): Maltodextrin for 28 days
  Interventions: Dietary Supplement: Maltodextrin placebo

INTERVENTIONS:
Dietary Supplement: Inulinase — Participants will consume one capsule containing 1,000 INU inulinase, twice daily, for 28 days. Participants will be directed to consume the capsules with their two largest meals.
  Other Names: Fructan hydrolyase; Beta-fructofuranosidase
  Arms: Inulinase
Dietary Supplement: Maltodextrin placebo — Participants will consume one capsule containing maltodextrin, twice daily, for 28 days. Participants will be directed to consume the capsules with their two largest meals.
  Arms: Placebo

SUMMARY:
The objectives of this clinical trial are to: 1) assess the effect of microbial inulinase on gastrointestinal symptoms in healthy participants compared to a placebo, and 2) to assess the safety and tolerability of microbial inulinase in healthy participants compared to a placebo.

DETAILED DESCRIPTION:
Dietary FODMAPs (fermentable oligosaccharides, disaccharides, monosaccharides, and polyols) can be digestively bothersome for certain fiber-intolerant individuals, as well as those with irritable bowel syndrome (Dionne et al.). Oral supplementation of microbial enzymes is a promising strategy to ameliorate gastrointestinal (GI) symptoms-such as bloating, abdominal discomfort, and gas-that are associated with food intolerances. Oral enzyme supplementation with fungal beta-galactosidase (lactase), fungal alpha-galactosidase, and a mixture of microbial and plant proteases have previously been clinically shown to effectively reduce GI symptoms associated with dairy, legume, and gluten consumption, respectively (Lin et al.; Di Stefano et al.; Ido et al.). While alpha-galactosidase effectively hydrolyzes galactan-type FODMAPs, there remains a need to target fructan-type FODMAPs. Preclinical data using an in vitro static GI digestion model showed that the microbial enzyme inulinase can effectively digest fructan-rich substrates (e.g., inulin from chicory root, garlic, and a high-fructan meal mash) better than control conditions under simulated gastric conditions (Guice et al., submitted).

The present study is a randomized, double-blind, placebo-controlled clinical trial to determine the safety and tolerability of microbial inulinase as a digestive enzyme supplement in healthy adults. This clinical trial will include 60 participants who are healthy adults between the ages of 20 to 60 and who regularly consume at least two meals daily. The study duration will be up to 62 days. This trial consists of one screening visit (Visit 1, Day -30 to -15), a baseline visit (Visit 2, Day 1), and an end-of-study visit (Visit 3, Day 29 ± 3).

To assess the effect of inulinase on GI-related symptoms, participants will fill out the paper Gastrointestinal Symptom Rating Scale (GSRS) on a weekly basis over the course of the study. The GSRS is a validated questionnaire containing 15 questions used to assess symptoms that are commonly associated with GI disorders (Machnicki et al.). All 15 questions are rated using a 7-point Likert scale, where higher ratings represent more discomfort. The GSRS score is determined by the score of five subscales: reflux, diarrhea, abdominal Pain, indigestion, and constipation. The reflux score will be calculated as an average score of questions 2 and 3. The diarrhea score will be calculated as an average score of questions 11,12, and 14. The abdominal pain score will be calculated as an average score of questions 1, 4, and 5. The indigestion score will be calculated as an average score of questions 6, 7, 8, and 9. The constipation score will be calculated as an average score of questions 10, 13, and 15. Each subscale score is the domain score. The average of all 5 domain scores will give the GSRS score. The GSRS score and 5 sub-scale (domain) scores will be used for analysis. The scores in Visit 2 will be treated as baseline, and change from baseline to Week 1, Week 2, Week 3, and Week 4 will be calculated, as well as the proportion of participants showing improved scores.

At screening Visit 1 (up to 30 days and no less than 15 days prior to the baseline visit), participants will arrive at the clinic in a fasting state (≥ 10 hours). After participants provide voluntary informed consent, the following information will be recorded, and procedures carried out:

* Collect demographic data (age, sex, ethnicity and race)
* Review medical/health history
* Review/record dietary and lifestyle habits
* Review/record use of concomitant treatments
* Review inclusion/exclusion criteria
* Take anthropometric measurements [height (screening only), weight) and vital signs [heart rate (HR) and blood pressure (BP)]
* Calculate body mass index (BMI; kg/m^2)
* Perform a brief symptom-based physical exam, if necessary
* Collect blood for hematology, clinical chemistry, lipid profile, and hemoglobin A1c (HbA1c)
* Dispense GSRS questionnaire for in-clinic completion
* Dispense GSRS questionnaire for at-home use
* Dispense study product (placebo only) and study diary

After confirming eligibility, from Day -14 to Day -1 (the day prior to baseline visit on Day 1), all participants will complete a 2-week run-in period where they will orally consume the placebo capsule twice daily with their usual two largest meals of the day (one capsule per meal) with the same two meals each day.

At baseline Visit 2 (Day 1), participants will arrive at the clinic in a fasting state (≥ 10 hours). The following visit procedures will occur:

* Collect and review any unused study product
* Review the study diary to assess compliance, concomitant treatments, medical conditions, and changes in health
* Review inclusion/exclusion criteria
* Review medical/health history
* Review any changes in dietary and lifestyle habits
* Take anthropometric measurements and vital signs (HR and BP)
* Calculate BMI using height collected from screening
* Collect blood for hematology, clinical chemistry, and lipid profiling
* Collect blood for lactate, insulin, uric acid, and high sensitivity C-reactive protein (hsCRP)
* Collect urine for pregnancy test
* Collect the GSRS questionnaire completed during the run-in period
* Dispense GSRS questionnaire for the participant to complete in-clinic
* Dispense GSRS questionnaire for at-home use
* Randomize the participant to inulinase or placebo
* Dose of study product in-clinic
* Adverse Event (AE) monitoring
* Dispense study products and study diary for home use by the participant

At the baseline visit on Day 1, participants will be randomized in a 1:1 ratio to either study product [1,000 units of inulinase activity (INU) per serving] or placebo and then start the 28 ± 3 days of twice daily study product consumption. Study product will be taken in the same manner (1 capsule taken twice daily with their two usual larger meals of the day).

At end-of-study Visit 3 (Day 29 ± 3), participants will arrive at the clinic in a fasting state (≥ 10 hours). The following visit procedures will occur:

* Return any unused study product and packaging of used study product
* Collect and review the study diary to assess compliance
* Review any changes in dietary and lifestyle habits
* Measure vital signs (BP and HR) and weight, and calculate BMI
* Collect urine for pregnancy test
* Collect blood for hematology, clinical chemistry, and lipid profiling
* Collect blood for lactate, insulin, uric acid, and hsCRP
* Collect the GSRS questionnaire and review for completion
* Dispense GSRS questionnaire for the participant to complete in-clinic
* AE monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult participants who are 20 to 60 years of age at screening (inclusive)
2. In good general health (no uncontrolled diseases or conditions) as deemed by the investigator and able to consume the study product
3. Regularly consumes at least 2 meals per day
4. Has a body mass index (BMI) between 18.5 to 29.9 kg/m^2 (inclusive) at Visit 2
5. Completes the run-in period with ≥ 90% product compliance for both consumption of doses and timing of doses as assessed by daily diary
6. Completes the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire during the run-in period
7. Individuals with childbearing potential must agree to practice an acceptable form of birth control for a certain time frame prior to the first dose of study product and throughout the study
8. Has maintained stable use of medication and supplements, and stable dietary and lifestyle habits, for the last 3 months prior to screening and agree to maintain them throughout the study
9. Agree to avoid strenuous exercise 24 hours prior to each visit
10. Willing to limit daily alcohol consumption to no more than 3-4 drinks per day throughout the study
11. Willing to maintain current use of cannabinoids (if applicable) throughout the study
12. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures

Exclusion Criteria:

1. Individuals who are lactating, pregnant, or planning to become pregnant during the study
2. Has a known sensitivity, intolerability, or allergy to any of the study products or their excipients
3. Received a vaccine for COVID-19 (coronavirus disease 2019) in the 2 weeks prior to screening or plans to receive a vaccine for COVID-19 during the study period, currently has COVID-19 or tests positive for COVID-19 within 28 days prior to baseline visit, or currently has any post COVID-19 condition(s) as defined by World Health Organization
4. Recent (within 2 weeks of Visit 1) history of an episode of acute gastrointestinal illness such as nausea, vomiting, or diarrhea
5. Have a history of irritable bowel syndrome, inflammatory bowel disease (including ulcerative colitis and Crohn's disease), functional constipation or diarrhea (defined by the Rome IV diagnostic criteria), celiac disease, malabsorption, gastroparesis, diverticulosis, gastric or duodenal ulcers, pancreatitis, or eating disorder; or have a history of intestinal surgery (excluding appendectomy or herniorrhaphy) or bariatric surgery.
6. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and/or digestion (e.g., history of bowel obstruction)
7. Participated in upper gastrointestinal endoscopy and/or colonoscopy or preparation within 3 months prior to Visit 1
8. Diagnosed with hypercholesterolemia or hypertriglyceridemia [i.e., elevated fasting low-density lipoprotein (LDL) (≥ 135 mg/dL; ≥ 3.5 mmol/L) or elevated triglycerides (≥ 150 mg/dL; ≥ 1.7 mmol/L) at screening]
9. Has a history of heart disease/cardiovascular disease, uncontrolled hypertension (≥ 140 systolic or ≥ 90 diastolic mmHg), kidney disease (dialysis or renal failure), hepatic impairment or disease
10. Is Type I or Type II diabetic or pre-diabetic [i.e., elevated fasting blood glucose levels (≥ 100 mg/dL; ≥ 5.6 mmol/L) and/or elevated hemoglobin A1c (≥ 6.0%) at screening]
11. Has a history of liver or gallbladder disease or stomach ulcers
12. Has a positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorders and/or immunocompromised
13. Diagnosed with cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit, or any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the results or the potential participant's ability to participate in the study
14. Major surgery in 3 months prior to screening or planned major surgery during the study
15. History of alcohol or substance abuse (including cannabinoids) in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program)
16. Extreme dietary habits at the discretion of the Qualified Investigator, evidenced by a diet wherein the ratio of individual macronutrients and dietary fiber is markedly different than the typical American diet [e.g., ketogenic diet, Atkins diet, low FODMAP (fermentable oligosaccharides, disaccharides, monosaccharides, and polyols) diet, vegetarian diet, fruitarian diet, etc.]
17. Use of any treatment listed in Study Protocol (No. B03-22-01-T0037) Section 6.5 (Concomitant Treatments) outside of the permitted time frames and/or conditions.
18. Receipt or use of investigational products in another research study within 28 days prior to baseline (Visit 2) or longer if the previous investigational product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study
19. Self-report of blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to screening or a blood donation of more than 450 mL within 56 days prior to baseline
20. Self-report of donating plasma (e.g., plasmapheresis) within 14 days prior to screening.
21. Any other active or unstable medical conditions or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale score | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 7, Day 14, Day 21, and Day 28 in Gastrointestinal Symptom Rating Scale scores (overall score and domain scores). All 15 questions are rated using a 7-point Likert scale (1 to 7), where lower ratings represent a better outcome or less discomfort.
Gastrointestinal Symptom Rating Scale improvement | 4 weeks
  Between placebo and inulinase treatments, percentage of participants showing improvement from baseline to Day 28 as assessed by reduction of Gastrointestinal Symptom Rating scores (overall score and domain scores). All 15 questions are rated using a 7-point Likert scale (1 to 7), where lower ratings represent a better outcome or less discomfort.
Abdominal discomfort, bloating, and burping scores | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 7, Day 14, Day 21, and Day 28 on individual Gastrointestinal Symptom Rating Scale questions on abdominal discomfort, bloating, and burping. These 3 questions are rated using a 7-point Likert scale (1 to 7), where lower ratings represent a better outcome or less discomfort.
Plasma lactate | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting plasma lactate concentration (mmol/L)
Serum insulin | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum insulin concentration (pmol/L)
Serum uric acid | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum uric acid concentration (umol/L)
Serum high-sensitivity C-reactive protein (hsCRP) | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum hsCRP concentration (mg/L)
Serum total cholesterol | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum total cholesterol concentration (mmol/L)
Serum low-density lipoprotein (LDL) cholesterol | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum LDL cholesterol concentration (mmol/L)
Serum high-density lipoprotein (HDL) cholesterol | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum HDL cholesterol concentration (mmol/L)
Plasma high-density lipoprotein (HDL) cholesterol | 6 weeks
  Between placebo and inulinase treatments, change from screening to Day 28 in fasting plasma HDL cholesterol concentration (mg/dL)
Serum triglycerides | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum triglycerides concentration (mmol/L)
Serum albumin | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum albumin concentration (g/L)
Serum alkaline phosphatase | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum alkaline phosphatase concentration (U/L)
Serum alanine transaminase | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum alanine transaminase concentration (U/L)
Serum aspartate transaminase | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum aspartate transaminase concentration (U/L)
Serum chloride | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum chloride concentration (mmol/L)
Serum creatinine | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum creatinine concentration (umol/L)
Serum globulin | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum globulin concentration (g/L)
Serum glucose | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum glucose concentration (mmol/L)
Serum potassium | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum potassium concentration (mmol/L)
Serum sodium | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum sodium concentration (mmol/L)
Serum total bilirubin | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum total bilirubin concentration (umol/L)
Serum total protein | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting serum total protein concentration (g/L)
Whole blood basophils | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood basophil count (x 10^9/L)
Whole blood eosinophils | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood eosinophil count (x 10^9/L)
Whole blood hematocrit | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood hematocrit (as volume percent)
Whole blood hemoglobin | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood hemoglobin concentration (g/dL)
Whole blood lymphocytes | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood lymphocyte count (x 10^9/L)
Whole blood mean corpuscular hemoglobin | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood mean corpuscular hemoglobin (pg)
Whole blood mean corpuscular hemoglobin concentration | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood mean corpuscular hemoglobin concentration (g/L)
Whole blood mean corpuscular volume | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood mean corpuscular volume (fL)
Whole blood monocytes | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood monocyte count (x 10^9/L)
Whole blood neutrophils | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood neutrophil count (x 10^9/L)
Whole blood platelets | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood platelet count (x 10^9/L)
Whole blood mean platelet volume | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood mean platelet volume (fL)
Whole blood red blood cells | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood red blood cell count (x 10^9/L)
Whole blood red blood cell distribution width | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood red blood cell distribution width
Whole blood white blood cells | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in fasting whole blood white blood cell count (x 10^9/L)
Whole blood hemoglobin A1c (HbA1c) | Day 1
  Fasting whole blood HbA1c concentration at Day 1 (%)
Estimated glomerular filtration (eGFR) | 4 weeks
  Between placebo and inulinase treatments, change from baseline to Day 28 in eGFR (mL/min/1.73m^2)
Blood pressure | 4 weeks
  Resting systolic blood pressure over resting diastolic blood pressure (mmHg/mmHg)
Heart rate | 4 weeks
  Resting heart rate (beats per minute)
Body weight | 4 weeks
  Body weight (kg)
Body mass index | 4 weeks
  Body mass index (kg/m^2)
Incidence of adverse events | 4 weeks
  Number of participants with adverse events
Incidence of serious adverse events | 4 weeks
  Number of participants with serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, CCFP, Principal Investigator — Apex Trials
Locations (1):
- Nutrasource site (Apex Trials), Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garvey SM, LeMoire A, Wang J, Lin L, Sharif B, Bier A, Boyd RC, Baisley J. Safety and Tolerability of Microbial Inulinase Supplementation in Healthy Adults: A Randomized, Placebo-Controlled Trial. Gastro Hep Adv. 2024 Jun 21;3(7):920-930. doi: 10.1016/j.gastha.2024.05.013. eCollection 2024. PMID 39318719
- [Background] Dionne J, Ford AC, Yuan Y, Chey WD, Lacy BE, Saito YA, Quigley EMM, Moayyedi P. A Systematic Review and Meta-Analysis Evaluating the Efficacy of a Gluten-Free Diet and a Low FODMAPs Diet in Treating Symptoms of Irritable Bowel Syndrome. Am J Gastroenterol. 2018 Sep;113(9):1290-1300. doi: 10.1038/s41395-018-0195-4. Epub 2018 Jul 26. PMID 30046155
- [Background] Lin MY, Dipalma JA, Martini MC, Gross CJ, Harlander SK, Savaiano DA. Comparative effects of exogenous lactase (beta-galactosidase) preparations on in vivo lactose digestion. Dig Dis Sci. 1993 Nov;38(11):2022-7. doi: 10.1007/BF01297079. PMID 8223076
- [Background] Di Stefano M, Miceli E, Gotti S, Missanelli A, Mazzocchi S, Corazza GR. The effect of oral alpha-galactosidase on intestinal gas production and gas-related symptoms. Dig Dis Sci. 2007 Jan;52(1):78-83. doi: 10.1007/s10620-006-9296-9. Epub 2006 Dec 7. PMID 17151807
- [Background] Ido H, Matsubara H, Kuroda M, Takahashi A, Kojima Y, Koikeda S, Sasaki M. Combination of Gluten-Digesting Enzymes Improved Symptoms of Non-Celiac Gluten Sensitivity: A Randomized Single-blind, Placebo-controlled Crossover Study. Clin Transl Gastroenterol. 2018 Sep 19;9(9):181. doi: 10.1038/s41424-018-0052-1. PMID 30228265
- [Background] Machnicki G, Pefaur J, Gaite L, Linchenco AM, Raimondi C, Schiavelli R, Otero A, Margolis MK. Gastrointestinal (GI)-Specific patient reported outcomes instruments differentiate between renal transplant patients with or without GI symptoms: results from a South American cohort. Health Qual Life Outcomes. 2008 Jul 21;6:53. doi: 10.1186/1477-7525-6-53. PMID 18644133